CLINICAL TRIAL: NCT06232213
Title: The PTC Microtumor Model is Used to Guide the Feasibility Study of Treatment for Patients With Drug-resistant or Relapsed Advanced Ovarian Epithelial Cancer or Endometrial Cancer
Brief Title: Clinical Study of Individualized Treatment of Relapsed or Drug-resistant Advanced Gynecological Tumors Guided by PTC Model
Status: Recruiting | Type: Observational
Sponsor: Hua Li (Other)
Responsible Party: Sponsor-Investigator, Hua Li, Department of Obstetrics and Gynecology, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Other Study IDs: LH2401
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Personalized Cancer Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: The results of PTC microtumor model were used to guide treatment, including 12 cases of ovarian cancer and 8 cases of endometrial cancer.
- control group: Patients who did not use the PTC model to guide treatment during the same period included 12 cases of ovarian cancer and 8 cases of endometrial cancer.

SUMMARY:
The clinical treatment of patients with resistant/relapsed/advanced gynecological malignancies is very difficult, and the difficulty lies in the selection of effective drugs. This study was a cohort study of recurrent/drug-resistant advanced ovarian high-grade serous carcinoma and advanced/recurrent endometrial adenocarcinoma treated in our hospital. A total of 20 cases were included in the proposed study group, including 12 cases of high-grade serous ovarian carcinoma and 8 cases of endometrial adenocarcinoma. Twenty patients who did not use PTC model to guide treatment at the same period were selected as controls. To compare the consistency of in vitro drug sensitivity detection results of PTC microtumor with clinical therapeutic effect, and to explore the feasibility of using PTC microtumor model to guide the treatment of patients with drug-resistant/recurrent advanced ovarian epithelial cancer or endometrial cancer. The clinical therapeutic effects of the study group and the control group were compared, and the rates of CR, PR, SD, PFS, OS and TTP were evaluated by RECIST1.1 standard. PTC models based on different clinical samples (tissue and ascites) were compared to analyze the consistency of in vitro drug sensitivity detection results and the relationship with clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, ≤80 years
2. Recurrent/drug-resistant gynecological tumors include: ① patients with advanced high-grade ovarian serous cancer whose tumor is uncontrolled or recurrent within 6 months after receiving platinum-based chemotherapy; ② Advanced ovarian high-grade serous cancer patients with platinum resistance at first treatment; ③ Patients with advanced or recurrent endometrial adenocarcinoma.
3. Life expectancy > 6 months;
4. Malignant tumors that are not being treated by other systems or are in an active phase;
5. Have at least one measurable target lesion according to RECIST1.1 criteria;
6. Specimen requirements: fresh specimens with sufficient cell culture, including tissue samples and abdominal effusion;
7. Physical strength score: ECOG 0-2;
8. Major organ functions must meet clinical treatment requirements:

   * Blood routine: neutrophil (ANC) ≥1.5x109/L; Platelet count (PLT) ≥90x109/L; Hemoglobin (Hb) ≥90g/L; ② Blood biochemistry: total bilirubin (TBIL) ≤1.5x upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5xULN; Urea nitrogen (BUN) and creatinine (Cr) ≤1.5 x ULN

(3) Heart color ultrasound: left ventricular ejection fraction (LVEF) ≥55%;

④ 12-lead ECG: Fridericia method corrected QT period (QTcF) < 470 msec. (9) Consent to abstinence from sex or use of an effective contraceptive method during treatment and for at least 7 months after the last dose in the study treatment for female patients who are not menopausal or have not been surgically sterilized; (10) Patients participating in the study (or their legal representatives) understand and voluntarily sign informed consent, have good compliance, and are willing to cooperate with follow-up.

Exclusion Criteria:

1. Patients who are unable to provide sufficient fresh samples;
2. pregnant and lactating women, female patients with fertility and positive pregnancy tests, or patients of childbearing age who are unwilling to take effective contraceptive measures during the whole test period;
3. The patient has uncontrollable co-morbidity, including but not limited to: symptomatic congestive heart failure, unstable angina pectoris and myocardial infarction, uncontrolled grade III hypertension, liver insufficiency, renal insufficiency, diabetes uncontrolled blood sugar, arrhythmia and mental illness;
4. Other circumstances in which the investigator determines that participation in the study is not appropriate.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recurrent/drug-resistant and advanced ovarian high-grade serous carcinoma and advanced/recurrent endometrial adenocarcinoma were treated at Beijing Chaoyang Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
tumor remission status | 24 months
  According to RECIST v1.1 criteria, patients were evaluated for tumor remission status (complete response (CR), partial response (PR), stable disease (PR), etc.). SD) or progressive disease (PD).

CONTACTS AND LOCATIONS:
Locations (1):
- Bei Jing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No